CLINICAL TRIAL: NCT03293927
Title: Investigating Polypharmacy-related Adverse Events in Critically Ill Children
Brief Title: Polypharmacy-related Adverse Events in Critically Ill Children
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled in study.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00084476
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2018-10

CONDITIONS: Delirium
Keywords: children, mechanically ventilated, fentanyl, dexmedetomidine, delirium, polypharmacy
MeSH Terms: conditions — Delirium | interventions — Fentanyl; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Fentanyl + Dexmedetomidine (Experimental)
  Interventions: Drug: Fentanyl; Drug: Dexmedetomidine
- Dexmedetomidine + Fentanyl (Experimental)
  Interventions: Drug: Fentanyl; Drug: Dexmedetomidine
- Fentanyl only (Experimental)
  Interventions: Drug: Fentanyl
- Dexmedetomidine only (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Fentanyl — The patient will receive IV fentanyl
  Arms: Dexmedetomidine + Fentanyl; Fentanyl + Dexmedetomidine; Fentanyl only
Drug: Dexmedetomidine — The patient will receive IV dexemedetomidine
  Arms: Dexmedetomidine + Fentanyl; Dexmedetomidine only; Fentanyl + Dexmedetomidine

SUMMARY:
The purpose of this study is to learn how 2 medications (fentanyl and dexmedetomidine) affect how sick children think and interact with their environments.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2-<18 at the time of enrollment
* Admitted to the Duke PICU or PCICU
* Planned or anticipated mechanically ventilation for ≥2 days
* Require sedation to maintain mechanical ventilation
* No contraindication to receipt of fentanyl or dexmedetomidine per clinician judgment
* Availability and willingness of the parent/legal guardian to provide written informed consent

Exclusion Criteria:

* Any concomitant condition, which in the opinion of the investigator would preclude a subject's participation in the study.
* Previous participation in this study
* Planned receipt of sedatives other than fentanyl or dexmedetomidine
* Participants with any of the following diagnoses: traumatic brain injury, intracranial hemorrhage, baseline neurodevelopmental delay, status epilepticus, or requiring inotropic support for hemodynamic stability.
* Renal failure requiring renal replacement therapy
* Hepatic failure
* Support with extracorporeal membrane oxygenation

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in delirium scores as measured by CAPD score | up to 10 days

SECONDARY OUTCOMES:
Drug level associated with CAPD score | up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Kanecia Zimmerman, MD, Principal Investigator — Duke
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States